CLINICAL TRIAL: NCT05942014
Title: Correlation of Children's Electronic Screen Time Exposure and Dental Anxiety and Behavior in a Group of Egyptian Children
Brief Title: Correlation of Children's Electronic Screen Time Exposure and Dental Anxiety and Behavior
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Ali Kadry Hassanen, doctor, Cairo University
Other Study IDs: dental anxiety and screen time
Record Dates: First submitted 2023-06-21; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Children's Screen Exposure
Keywords: dental anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: dental anxiety — Evaluate dental anxiety in children and its relation with screen time exposure
  Other Names: screen time exposure

SUMMARY:
This study aims to detect the correlation between children's electronic screen time exposure and dental anxiety and behavior in a group of Egyptian children

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 6-to-8-years old
* First dental visit
* Both genders

Exclusion Criteria:

* Children with Mental or neurological disorders.
* Children with Systemic disorders.
* Children who use medications that could interfere with the central nervous system
* Children with previous hospitalization

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All medically free male and female Egyptian children with age from 6 to 8 years that have a first dental visit
Sampling Method: Non-Probability Sample
Enrollment: 211 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Child dental anxiety | "through study completion, an average of 1 year"
  Abeer children dental anxiety SCALE,Questionnaire
Assessment of the child's behavior during the dental visit | "through study completion, an average of 1 year"
  Frankl Behavioral Rating Scale,Questionnaire

SECONDARY OUTCOMES:
Exposure to electronic screens | "through study completion, an average of 1 year"
  Questionnaire

REFERENCES:
- [Result] Mobarek NH, Khalil AM, Talaat DM. Exposure to Electronic Screens and Children's Anxiety and Behavior During Dental Treatment. J Dent Child (Chic). 2019 Sep 15;86(3):139-144. PMID 31645254
- [Result] Alaki SM, Al-Raddadi RA, Sabbagh HJ. Children's electronic screen time exposure and its relationship to dental anxiety and behavior. J Taibah Univ Med Sci. 2023 Jan 10;18(4):778-786. doi: 10.1016/j.jtumed.2022.12.021. eCollection 2023 Aug. PMID 36852238